CLINICAL TRIAL: NCT06819059
Title: Safety and Efficacy of Pediatric Cardiac Telerehabilitation in Adolescents With Heart Disease
Brief Title: Safety and Effectiveness of a Virtual Pediatric Cardiac Rehabilitation Program or Telerehabilitation in Children With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Aimee Layton, Associate Professor of Applied Physiology in Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAT7872
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Congenital Abnormalities; Pulmonary Arterial Hypertension (PAH); Orthotopic Heart Transplant; Cardiac Rehabilitation; Pediatric Cardiology; Telehealth; Telerehabilitation
Keywords: Pediatric Cardiac Telerehabilitation; Pediatric Exercise; Cardiac Rehabilitation
MeSH Terms: conditions — Congenital Abnormalities; Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, with optional cross over for control participants to receive the treatment after completing 3 months of control data collection and post 3 month enrollment follow up testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 is the treatment arm that receives 12 weeks of weekly cardiac telerehabilitation sessions (Experimental): The participants randomized to study Arm 1 were enrolled in the 12 weeks of cardiac telerehabilitation which included weekly one-on-one sessions with the exercise physiologist or physical therapist. Participants in this arm also received fitness activity trackers to record heart rate, active minutes, steps and sleep data.
  Interventions: Behavioral: Pediatric Cardiac Telerehabilitation; Behavioral: Fitness Tracker Only
- Arm 2 was the study arm for participants randomized to the control group (Active Comparator): Participants randomized to Arm 2 received fitness activity trackers that provided the patient with heart rate data, steps and sleep data but received no formal exercise training.
  Interventions: Behavioral: Fitness Tracker Only

INTERVENTIONS:
Behavioral: Pediatric Cardiac Telerehabilitation — The program was entirely virtual except for pre and post program cardiopulmonary exercise testing. Patients were provided a stationary bicycle, hand weights, and resistance training bands. They exercised over zoom with a physical therapist or exercise physiologist weekly and were also asked to exercise independently 2x per week. Electrocardiograms (ECGs) were provided to the patients as a single lead monitor and results were shared with the study team after each session or during sessions if the patient reported symptoms. Compliance and activity data were recorded using Fitbit activity trackers.
  Arms: Arm 1 is the treatment arm that receives 12 weeks of weekly cardiac telerehabilitation sessions
Behavioral: Fitness Tracker Only — Control participants were provided fitness trackers and weekly text messaging from the study team to synch their devises but no formal exercise training. They were allowed to enroll in the exercise training after completing 3 months as a control.

SUMMARY:
Cardiac telerehabilitation is a much-needed pediatric therapy; however, a lack of randomized controlled trials has limited the development of and reimbursement for this valuable service. Through this prospective, randomized controlled trial, the investigators aim to demonstrate the safety and efficacy of PCTR in a clinically diverse population of children and adolescents with heart disease.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized, controlled pilot of a pediatric cardiac telerehabilitation program in adolescents with acquired or congenital heart disease.

Because of the known benefits of exercise, controls were offered the opportunity to participate in the intervention group after completing the 12 weeks in the control group.

Participants were randomized in a 2:1 ratio (intervention: control) to maximize participation in the exercise intervention. Participants were from three core populations: primary or secondary pulmonary hypertension (PH), structural congenital heart disease (CHD), and post-orthotopic heart transplant (OHT). PCTR was "semi-supervised", where one day per week the participant exercised one-on-one with a physical therapist or exercise physiologist via virtual platform and 2 days per week they exercised independently. Participants wore an activity tracker with heart rate monitoring 24 hours a day and a single lead, chest-based electrocardiogram (ECG) device while exercising. A physician or program director reviewed ECGs after all sessions. An adult had to be available in case of an emergency during each session. Controls received weekly check-ins and a Fitbit but did not receive a formal exercise prescription. All participants underwent baseline and post-study assessments including the cardiopulmonary stress test (CPET) and questionnaires and wore their Fitbits for the duration of the study.

Compliance was measured by attendance of Zoom appointments, Fitbit activity data, Wellue single lead electrocardiogram (ECG) data, and self-reported activity performed. Efficacy was measured by CPET results, validated questionnaire data and activity levels as determined by Fitbit data.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 -25 yrs
* Not participating in organized sports of physical fitness programs
* Able to follow basic directions and express symptoms
* Dx of pulmonary hypertension, congenital heart disease, and transplant programs
* Clinically stable as deemed by the referring cardiologist

Exclusion Criteria:

* Clinical instability as demonstrated by recent medication escalation (within 3 months prior to starting the program)
* Hemodynamic instability
* Significant arrhythmia or ST segment or T wave abnormalities
* End-tidal carbon dioxide less than 20 mmHg with exercise, or exercise-induced symptoms that would limit ability to participate in the intervention safely

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Sessions Completed | 12 weeks
  The primary outcome of this study was compliance measured by drop out rate of the cardiac rehabilitation group and any adverse events that occurred with exercise.

SECONDARY OUTCOMES:
Change in exercise time | 12 weeks
  The study will measure the change in exercise duration pre- to post-intervention.
Change in Anxiety associated with exercise (ESQ -18) | 12 weeks
  The impact on anxiety associated with exercise before and after the program will be measured using the Exercise Sensitivity Questionnaire on a 0-72 scale. Lower score indicates better outcome.
Change in Disease Burden by lower Quality of Life Measure | 12 weeks
  The impact of disease burden on quality of life using the PedsQL questionnaire (Pediatric Quality of Life) with a 0-60 scale, with a lower score indicating a lesser impact.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee M Layton, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - New York Presbyterian's Morgan Stanley's Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We would need clearance from our institutions legal services.